CLINICAL TRIAL: NCT02137681
Title: 2 Cycles Rituximab Compared With Standard Regimen in Management of ITP
Brief Title: A Multicentre Investigation of 2 Cycles Rituximab Compared With Standard Regimen in Management of Steroid-Resistant/Relapsed Immune Thrombocytopenia （ITP）
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No eligible patient was enrolled.
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITP-RTX2vs4
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2014-05

CONDITIONS: Immune Thrombocytopenia
Keywords: immune thrombocytopenia; rituximab; efficacy; safety
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 cycles (Experimental): 2 cycles RTX
  Interventions: Drug: Rituximab
- standard 4 cycles (Active Comparator): standard 4 cycles RTX
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab was given intravenously at a dose of 375mg/m(2) weekly for 2 consecutive weeks (Day 1, 8) in 2 cycles arm; or 4 consecutive weeks (Day 1, 8, 15, 22) in standard 4 cycles arm

SUMMARY:
The project was undertaking by Qilu Hospital, Shandong University and other several well-known hospitals in China. In order to report the efficacy and safety of Rituximab in different frequencies for the treatment of adults with steroid-resistant/relapsed immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
The investigators are undertaking a parallel group, multicentre, randomised controlled trial of 60 refractory ITP adult patients from medical centers in China. One part of the participants are randomly selected to receive rituximab (given intravenously at a dose of 375mg/m(2) weekly for 2 weeks, i.e. Day 1, 8; the others are selected to receive standard rituximab treatment (given intravenously at a dose of 375 mg/m(2) weekly for 4 cycles, i.e. Day 1, 8, 15, 22). Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study. In order to report the efficacy and safety of the combination therapy compared to conventional rituximab therapy for the treatment of adults with steroid-resistant/relapsed immune thrombocytopenia (ITP).

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for immune thrombocytopenia.
2. Untreated hospitalized patients, may be male or female, between the ages of 18 ~ 80 years.
3. To show a platelet count <30×10^9/L, and with bleeding manifestations.
4. Willing and able to sign written informed consent.

Exclusion Criteria:

1. Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 3 months before the screening visit.
2. Received second-line ITP-specific treatments (eg, cyclophosphamide, 6-mercaptopurine, vincristine, vinblastine, etc) within 3 months before the screening visit.
3. Received high-dose steroids or IVIG in the 3 weeks prior to the start of the study.
4. Current HIV infection or hepatitis B virus or hepatitis C virus infections.
5. Severe medical condition (lung, hepatic or renal disorder) other than chronic ITP. Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia)
6. Female patients who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period.
7. Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test.
8. Patients who are deemed unsuitable for the study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Early Response | 3 months
  response rate (CR+R) at the 3rd month from the initial injection of RTX. CR is defined as platelet count ≥ 100×10^9/L, and R is defined as platelet count of >30 × 10^9/L with a least a doubling of the baseline value.
Duration Response | 12 months
  response rate (CR+R) at the 12st month from the initial injection of RTX. CR is defined as platelet count ≥ 100×10^9/L, and R is defined as platelet count of >30 × 10^9/L with a least a doubling of the baseline value.

SECONDARY OUTCOMES:
Safety | 1 months
  The type and frequency of therapy associated adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, Dr., Principal Investigator — Shandong University
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China